CLINICAL TRIAL: NCT04523870
Title: Acute Effects of a Botanical Extract and Its Main Volatile Compound on Stress Response in Healthy Adults: Randomized, Cross-over (Three Arms), Double-blind, Placebo-controlled Clinical Trial
Brief Title: Acute Effects of a Botanical Extract and Its Main Volatile Compound on Stress Response in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Activ'inside (Industry)
Collaborators: CIC SANPSY (USR CNRS 3413), Groupe Hospitalier Pellegrin, Bordeaux, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: SAFRAI2018
Record Dates: First submitted 2020-07-30; First posted 2020-08-24 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Botanical extract (Experimental)
  Interventions: Dietary Supplement: Botanical extract
- Major compound of the extract (Experimental)
  Interventions: Dietary Supplement: Main compound of the botanical extract
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Botanical extract — One capsule
  Arms: Botanical extract
Dietary Supplement: Main compound of the botanical extract — one capsule
  Arms: Major compound of the extract
Dietary Supplement: Placebo — Maltodextrin, one capsule
  Arms: Placebo

SUMMARY:
The prevalence of stress in daily human life increase in the investigator's modern life style. Short stress, could be benefit for memory, but prolonged stress may conduct to disturbance in cardiovascular, neuroendocrine and central nervous systems. Moreover, it is well established that stress is the most common risk factor for the development of mood and anxiety disorders, such as major depressive disorder (MDD) and generalized anxiety disorder. In response to stress, hypothalamic-pituitary-adrenocortical (HPA) axis is one of activated pathway, which induce the cortisol release. Certain natural products could increase resilience to stress. Indeed, several preclinical studies have already showed that botanical extracts inhibited the typical plasmatic corticosterone elevation induced by an acute stress challenge. Therefore, the aim of this clinical trial is to investigate the acute effects of a botanical extract and one of his major compound, both delivered as sublingual single dose, on cortisol level, cardiac parameters, and psychometric response, in healthy adults exposed to an acute psychological stress.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker since at least 3 months
* Body Mass Index (BMI) in the normal range: 18.5 ≤ BMI < 25 kg/ m2 or "normal corpulence" according to investigator's judgment
* Usual waking hour between 6.00 and 9.00 am on weekdays
* Displaying a pattern of "reactive responder" to the stressor
* Subjects affiliated with a social security scheme
* Subjects capable of and willing to comply with the protocol and to give their written informed consent

Exclusion Criteria:

* Currently suffering from mental disorder or with personal history of such disease (depression, generalized anxiety disorder, obsessive compulsive disorder, panic disorder, simple phobia and social phobia, schizophrenia, …) according to the volunteer's self-declaration.
* Anxiolytic, antidepressant or any other treatment likely to affect some of the study parameters, whatever the reason of its prescription within the previous 3 months.
* Event (personal or professional) likely to have impacted the study parameters within 2 weeks before V1 (for example but not restricted to: change of professional function/ situation, death of a family member, divorce, surgery, accident, travel with jet lag …).
* Event (personal or professional) likely to affect the study parameters planned within the next 11 weeks, including but not restricted to: vaccination, travel with jet lag, …
* Systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg during the V0 visit (Blood pressure will be measured while the subject sit in a chair. Blood pressure will be measured after a 10-minute rest and will be repeated 3 times separated by 3-minute intervals. The average of the 3 measurements will be calculated.)
* Subjects diagnosed with at least one of the following will not be eligible:
* Present or recurrent infectious diseases (including cystitis, gingivitis, conjunctivitis, respiratory infections, …)
* Diabetes (type I or type II)
* Cardiovascular or vascular disease or history of cardiovascular or vascular disease (such as thrombosis, phlebitis, CVA, heart disease)
* Chronic disease affecting blood flow (examples: Raynaud's disease or syndrome, chronic veinous insuficiency)
* Allergic disease (asthma, allergic rhinitis, atopic dermatitis, …) or chronic inflammatory pathology (tendinitis, Crohn's disease, coeliac disease, …)
* Any other pathology which, according to investigator's judgment, is likely to affect the study parameters.
* Usual corticoïd treatment/ steroidal anti-inflammatory treatment (ex: Bétaméthasone, Cortivazol, Dexamethasone, Methylprednisolone, Prednisolone, Prednisone, Tétracosactide, Triamcinolone, …) including local treatments (ex : Locoïd lotion, Locatop, Locapred, Tridesonit, etc). Subjects will not be eligible if they have consumed such treatments within 2 weeks before V1 and/ or if they are likely to consume such treatments during the study;
* Oral antibiotic treatment within the last 2 weeks before entry into the study. In case of oral antibiotic started after inclusion, the next study visits of the participant will be reported until at least 2 weeks after the end of the antibiotic treatment.
* Unbalanced thyroid disease. However, subjects with controlled thyroid diseases (medication unchanged within the last 3 months) can be included;
* Suffering from a severe chronic pathology which, according to Investigator's judgment, is likely to affect at least one of the study parameters (such as but not restricted to: severe chronic pain, cancer or history of cancer unless in remission for more than 5 years, HIV, hepatitis, renal disease, cardiac disease);
* High physical activity practice: more than 10 hours per week of moderate to vigorous physical activity, or physical activity practice modified since less than 2 months or likely to be significantly modified within the next 11 weeks. Examples of moderate physical activity are: transporting light loads, bicycling at a normal pace, a double tennis, ... Walking is not considered as physical activity of moderate intensity.
* Subjects working in shift schedules (ex : nurse, baker, etc)
* Subjects whose working conditions are variable and likely to be extreme (ex: work in a cold room);
* Subjects consuming more than 3 coffee servings from waking until lunch (included), i.e. more than a bowl at breakfast + a cup in the morning + a cup at lunch.
* Subjects consuming any food supplement (including vitamins, minerals and botanicals and/or other substances) and refusing to stop for at least 2 weeks before V1 (inclusion visit) and until the end of his study participation;
* Usual alcohol consumption > 3 glasses/ day or chronic alcohol abuse treated since less than 3 months;
* Subjects with usual consumption of recreational drug. Subjects with occasional consumption of recreational drug can be include if they agree not to consume such products for at least one week before V1 and until the end of their study participation.
* Change in dietary habits since less than 4 weeks or planned within the next 11 weeks.
* Eating disorders: anorexia and bulimia or unstable dietary pattern.
* Any food allergy documented or suspected to one of the components of the study products.
* Subject presenting a psychological or linguistic inability to sign the informed consent.
* Subject under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision.
* Subject having received indemnities for clinical trial reaching at least 4500 Euros considering the last 12 months.
* Subject participating in another biomedical study or during the exclusion period of a previous study.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Cortisol response to an acute stress | Between baseline (before exposure to the stressor) and time 60 minutes after exposure to the stressor
  Area under the curve of the salivary cortisol concentration

SECONDARY OUTCOMES:
Maximum salivary cortisol concentration | Between baseline (before exposure to the stressor) and time 60 minutes after exposure to the stressor
Time of maximum of salivary cortisol concentration | Between baseline (before exposure to the stressor) and time 60 minutes after exposure to the stressor
Maximum change in heart rate variability parameters | Between baseline (before exposure to the stressor) and time 60 minutes after exposure to the stressor
Area under the curve of heart rate variability parameters | Between baseline (before exposure to the stressor) and time 60 minutes after exposure to the stressor
Maximum increase in the anxiety score | Between baseline (before exposure to the stressor) and time 60 minutes after exposure to the stressor
Time of maximum increase in the anxiety score | Between baseline (before exposure to the stressor) and time 60 minutes after exposure to the stressor
Area under the curve of the anxiety score | Between baseline (before exposure to the stressor) and time 60 minutes after exposure to the stressor
Maximum increase in the perceived stress score | Between baseline (before exposure to the stressor) and time 60 minutes after exposure to the stressor
Time of maximum increase in the perceived stress score | Between baseline (before exposure to the stressor) and time 60 minutes after exposure to the stressor
Area under the curve of the perceived stress score | Between baseline (before exposure to the stressor) and time 60 minutes after exposure to the stressor
Percentage of correct answers in serial subtractions | During the subtractions tasks
Percentage of correct answers given during stress test | During the 60 minutes of the stress test
Mean number of total answers given per second. | During the 60 minutes of the stress test

CONTACTS AND LOCATIONS:
Locations (1):
- SANPSY (CHU Pellegrin), Bordeaux, France